CLINICAL TRIAL: NCT01665755
Title: A Multicenter Randomised Controlled Trial Comparing Shock Success With Synchronized Defibrillation (Compression Upstroke Versus Precompression) During Ongoing Mechanical Cardiopulmonary Resuscitation In The Emergency Department
Brief Title: To Determine Optimal Time for Delivering Electrical Shocks to Cardiac Arrest Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Singapore General Hospital (Other)
Collaborators: Zoll Medical Corporation (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2011/456/C
Record Dates: First submitted 2012-08-06; First posted 2012-08-15 (Estimated); Last update posted 2019-09-20 (Actual); Status verified 2019-09

CONDITIONS: Cardiac Event; Sudden Cardiac Death; Death; Ventricular Fibrillation; Ventricular Tachycardia
MeSH Terms: conditions — Cardiovascular Diseases; Death, Sudden, Cardiac; Death; Ventricular Fibrillation; Tachycardia, Ventricular

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Precompression (Experimental): Control arm
  Interventions: Device: Precompression Defibrillation
- Upstroke Compression (Active Comparator): Intervention arm
  Interventions: Device: Upstroke Compression Defibrillation

INTERVENTIONS:
Device: Upstroke Compression Defibrillation
  Arms: Upstroke Compression
Device: Precompression Defibrillation
  Arms: Precompression

SUMMARY:
In this study, we are comparing the difference in outcomes between patients who were given shocks to the heart, during the upstroke of cardiopulmonary resuscitation (CPR) and before CPR is started. The study population will be all cardiac arrest patients attended by the staff of the Emergency Department who fulfil the eligibility criteria. Patients will be managed according to currently approved cardiac arrest protocols. Patients confirmed in cardiac arrest have manual chest compressions started while mechanical CPR (whereby chest compressions are delivered by an automated device) is prepared. Mechanical CPR should be started as soon as possible (<1 minute). If patients are eligible to be shocked, they will receive shocks either during upstroke of CPR or before CPR is started.

Thus the purpose of this study is to answer the question whether are there improvement in survival between when shocks are given during upstroke and before CPR is started.

DETAILED DESCRIPTION:
The purpose of this study will be to compare shock success during defibrillation synchronized with the upstroke of chest compression (peak upstroke), and precompression (control). This will be the world's first study to characterize the phase dependency of defibrillation during mechanical CPR in humans and to evaluate if optimal synchronized defibrillation can improve clinical outcomes.

The null hypothesis would be that there is no difference in shock success during defibrillation synchronized with the upstroke of chest compression (peak upstroke), and precompression (control). We will conduct statistical comparisons for the primary and secondary outcomes between the arms of the study.

The study population will be all cardiac arrest patients attended by the staff of the ED over the study period who fulfill the eligibility criteria. Patients will be managed according to currently approved cardiac arrest protocols. Patients confirmed in cardiac arrest with have manual chest compressions started while mechanical CPR is prepared. Mechanical CPR should be started as soon as possible (<1 minunte). If a shockable rhythm is present (VF/VT), patients will receive one of pre-randomized defibrillation protocols:

1. Synchronised defibrillation at peak-upstroke
2. Synchronised defibrillation at precompression

Definition of outcomes

* Shock success is defined as the termination of Ventricular Fibrillation (VF) or pulseless Ventricular Tachycardia (VT) and the establishment of organized rhythm within 60 seconds. An organized rhythm requires at least 2 QRS complexes separated by no more than 5 seconds.
* Survival to hospital discharge is defined as patient surviving the primary event and discharged from the hospital alive.
* Return of spontaneous circulation is defined as the presence of any palpable pulse, which is detected by manual palpation of a major artery.
* Survival to admission is defined as the admission to hospital without ongoing CPR or other artificial circulatory support.

ELIGIBILITY:
Inclusion Criteria:

* Cardiac Arrest patients who received eith CPR and/or defibrillation
* Ventricular Fibrillation or Pulseless Ventricular Tachycardia

Exclusion Criteria:

* Patients pronounced dead without attempting CPR according to standard operating procedure and ILCOR guidelines
* Cardiac arrest obviously caused by major trauma
* Children below age 21
* Patients who are pregnant

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 180 (Actual)
Dates: Start 2016-01 (Actual); Primary Completion 2018-03 (Actual); Study Completion 2019-04-03 (Actual)

PRIMARY OUTCOMES:
successful electrical conversion (shock success) | establishment of organized rhythm within 60 seconds
  Termination of Ventricular Fibrillation (VF) or pulseless Ventricular Tachycardia (VT) and the establishment of organized rhythm within 60 seconds. An organized rhythm requires at least 2 QRS complexes separated by no more than 5 seconds.

SECONDARY OUTCOMES:
termination of VF regardless of the resulting rhythm | at least 5 seconds after the shock
Return of spontaneous circulation (ROSC) | at least 20 minutes
Survival to hospital admission | at least 1 day
Survival to hospital discharge | at least 1 day
Functional survival outcomes assessed by the Glasgow Outcomes Score (CPC/OPC) | at least 1 day
European Quality of Life in 5 Dimensions | at least 1 day

CONTACTS AND LOCATIONS:
Overall Officials: Marcus Eng Hock Ong, MBBS, FRCS, Principal Investigator — Singapore General Hospital
Locations (1):
- Singapore General Hospital, Singapore, Singapore